CLINICAL TRIAL: NCT02416492
Title: A Double-Blind, Controlled Phase 2 Study of the Safety and Efficacy of Modified Stem Cells (SB623) in Patients With Chronic Motor Deficit From Traumatic Brain Injury (TBI)
Brief Title: A Study of Modified Stem Cells in Traumatic Brain Injury (TBI)
Acronym: STEMTRA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SanBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TBI-01
Record Dates: First submitted 2015-04-06; First posted 2015-04-15 (Estimated); Results first posted 2021-12-27 (Actual); Last update posted 2021-12-27 (Actual); Status verified 2021-11

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SB623 Cells (Experimental): SB623 Cells: 2.5, 5 or 10 million cells
  Interventions: Biological: SB623 cells
- Sham Surgery (Sham Comparator): Control Sham Surgery
  Interventions: Procedure: Sham Control

INTERVENTIONS:
Biological: SB623 cells — SB623 cells will be implanted in the peri-infarct area using stereotactic surgery.
  Arms: SB623 Cells
Procedure: Sham Control — Sham Surgery
  Arms: Sham Surgery

SUMMARY:
The primary purpose of the clinical study is to evaluate the clinical efficacy of intracranial administration of SB623 cells on patients with chronic motor deficit from Traumatic Brain Injury. A secondary purpose of the study is 1) to evaluate the effect of intracranial administration of SB623 cells on disability parameters and 2) to evaluate the safety and tolerability of intracranial administration of SB623 cells. Patients with stable, chronic motor deficits secondary to focal traumatic brain injury must be 12 months post TBI.

DETAILED DESCRIPTION:
This study was a multicenter, randomized (3:1) double-blind, active and sham-surgery controlled study to evaluate the safety, tolerability, and efficacy of stereotactic intracranial injection of SB623 cells in patients with fixed motor deficits from TBI. The study was conducted at approximately 22 sites across the United States, Ukraine, and Japan.

Two groups, Group 1 and Group 2, received investigational product SB623 and sham surgery, respectively, in a 3:1 randomization scheme. Group 1 was further randomized in a 1:1:1 ratio to receive either 2.5 million, 5 million, or 10 million SB623 cells. Randomization was performed via an interactive web response system (IWRS).

ELIGIBILITY:
Inclusion Criteria:

* Documented history of TBI, with correlated MRI or CT
* At least 12 months post-TBI
* Focal cerebral injury able to be identified on MRI (+/- concomitant diffuse axonal injury)
* Neurological motor deficit substantially due to focal cerebral injury observed on MRI
* GOS-E score of 3-6 (i.e. moderate or severe disability)
* Require Motricity Index 10-81 (UE Scale) and/or 10-78 (LE Scale)
* Able and willing to undergo computed tomography (CT) and magnetic resonance imaging (MRI)
* Subjects must be willing to participate in study related exercises to the extent possible
* Able to undergo all planned neurological assessments

Exclusion Criteria:

* History or presence of any other major neurological disease
* Any seizures in the prior 3 months
* The presence of contracture at any joints that would interfere with interpretation of any of the neurological assessments (e.g. contracture preventing the detection of any increase in the range of motion or ability to perform a task)
* Other neurologic, neuromuscular or orthopedic disease that limits motor function
* Clincially significant finding on MRI of brain not related to TBI
* Known presence of any malignancy except squamous or basal cell carcinoma of the skin
* History of CNS malignancy
* Positive findings on tests for occult malignancy, unless a non-malignant etiology is confirmed
* Uncontrolled systemic illness, including, but not limited to: hypertension (systolic >150 mm Hg or diastolic >95 mm Hg); diabetes; renal, hepatic, or cardiac failure
* Uncontrolled major psychiatric illness, including depression symptoms (CESD-R Scale of ≥16)
* Unexplained abnormal preoperative test values (blood tests, electrocardiogram [ECG], chest X-ray); x-ray evidence of infection; uncontrolled atrial fibrillation or uncontrolled congestive heart failure
* Presence of craniectomy (without bone flap replacement) or other contraindication to stereotactic surgery
* Participation in any other investigational trial within 4 weeks of initial screening or within 7 weeks of study entry
* Botulinum toxin injection, phenol injection, intrathecal baclofen, or any other interventional treatments for spasticity (except bracing and splinting) 16 weeks priot to the Baseline visit.
* Ongoing use of other non-traditional drugs
* Substance use disorder (per DSM-V criteria, including drug or alcohol)
* Contraindications to head CT or MRI
* Pregnant or lactating
* Female patients of childbearing potential unwilling to use an adequate birth control method during the 12 months of the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2016-07-06 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-03-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel C Lu, MD, PhD, Principal Investigator — University of California, Los Angeles, Department of Neurosurgery
Locations (36):
- United States (25):
  - UCLA Medical Center (Surgical/Assessment), Los Angeles, California
  - Ronald Reagan UCLA Medical Denter, Los Angeles, California
  - The Research Center of Southern California, LLC (Assessment), Oceanside, California
  - University of California, Irvine (Assessment/Surgical), Orange, California
  - Westview Clinical Research (Assessment), Placentia, California
  - Providence Saint John's Health Center, Santa Monica, California
  - John Wayne Cancer Institute at Providence St. Johns Health Center, Santa Monica, California
  - Stanford Health Care (Surgical/Assessment), Stanford, California
  - Craig Hospital, Englewood, Colorado
  - Ki Health Partners, LLC dba New England Institute for Clinical Research (Assessment), Stamford, Connecticut
  - SouthCoast Research Center, Miami, Florida
  - Midtown Neurology, PC (Assessment), Atlanta, Georgia
  - Emory University Hospital (Surgical), Atlanta, Georgia
  - Rehabilitation Institute of Chicago, Chicago, Illinois
  - Shirley Ryan Ability Lab, Chicago, Illinois
  - NYU Langone Medical Center (Surgical/Assessment), New York, New York
  - New York University Langone Medical Center, New York, New York
  - Burke Rehab Center (Assessment), White Plains, New York
  - Ohio Health Research, Columbus, Ohio
  - Moss Rehab (Assessment), Elkins Park, Pennsylvania
  - University of Pittsburgh Medical Center (Surgical/Assessment), Pittsburgh, Pennsylvania
  - University of Pittsburgh School of Medicine, Pittsburgh, Pennsylvania
  - Medical University of South Carolina (Surgical), Charleston, South Carolina
  - Virginia Commonwealth University, Richmond, Virginia
  - Mid-Columbia Research, Richland, Washington
- Japan (10):
  - Hokkaido University Hospital (Surgical/Assessment), Sapporo, Hokkaido
  - Yokohama City University Hospital (Surgical/Assessment), Yokohama, Kanagawa
  - Okayama University Hospital (Assessment/Surgical), Okayama, Okayama-ken
  - Osaka University Hospital (Assessment/Surgical), Suita, Osaka
  - University of Tokyo Hospital (Assessment/Surgical), Bunkyo, Tokyo
  - Hokkaido University Hospital, Hokkaido
  - Okayama University Hospital, Okayama
  - Osaka University Hospital, Osaka
  - University of Tokyo Hospital, Tokyo
  - Yokohama City University Hospital, Yokohama
- Clinical Hospital Feofaniia, Kiev, Ukraine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Okonkwo DO, McAllister P, Achrol AS, Karasawa Y, Kawabori M, Cramer SC, Lai A, Kesari S, Frishberg BM, Groysman LI, Kim AS, Schwartz NE, Chen JW, Imai H, Yasuhara T, Chida D, Nejadnik B, Bates D, Stonehouse AH, Richardson RM, Steinberg GK, Poggio EC, Weintraub AH. Mesenchymal Stromal Cell Implants for Chronic Motor Deficits After Traumatic Brain Injury: Post Hoc Analysis of a Randomized Trial. Neurology. 2024 Oct 8;103(7):e209797. doi: 10.1212/WNL.0000000000209797. Epub 2024 Sep 4. PMID 39231380
- [Derived] McCrea MA, Cramer SC, Okonkwo DO, Mattke S, Paadre S, Bates D, Nejadnik B, Giacino JT. Determining minimally clinically important differences for outcome measures in patients with chronic motor deficits secondary to traumatic brain injury. Expert Rev Neurother. 2021 Sep;21(9):1051-1058. doi: 10.1080/14737175.2021.1968299. Epub 2021 Aug 26. PMID 34402352
- [Derived] Kawabori M, Weintraub AH, Imai H, Zinkevych I, McAllister P, Steinberg GK, Frishberg BM, Yasuhara T, Chen JW, Cramer SC, Achrol AS, Schwartz NE, Suenaga J, Lu DC, Semeniv I, Nakamura H, Kondziolka D, Chida D, Kaneko T, Karasawa Y, Paadre S, Nejadnik B, Bates D, Stonehouse AH, Richardson RM, Okonkwo DO. Cell Therapy for Chronic TBI: Interim Analysis of the Randomized Controlled STEMTRA Trial. Neurology. 2021 Feb 22;96(8):e1202-e1214. doi: 10.1212/WNL.0000000000011450. PMID 33397772

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Group: SB623 2.5 Million Cells: 2.5 million SB623 cells
  SB623 surgically implanted
- Treatment Group: SB623 5 Million Cells: 5 million SB623 cells
  SB623 surgically implanted
- Treatment Group: SB623 10 Million Cells: 10 million SB623 cells
  SB623 surgically implanted
- Treatment Group: Sham Surgery: Control Sham Surgery
  Sham Control: Sham Surgery
Period: Overall Study
Arm/Group | Treatment Group: SB623 2.5 Million Cells | Treatment Group: SB623 5 Million Cells | Treatment Group: SB623 10 Million Cells | Treatment Group: Sham Surgery
Started | 15 | 15 | 16 | 15
Completed | 15 | 15 | 16 | 15
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment Group: 2.5 Million Cells: 2.5 million SB623 cells
  SB623 surgically implanted
- Treatment Group: 5 Million Cells: 5 million SB623 cells
  SB623 surgically implanted
- Treatment Group: 10 Million Cells: 10 million SB623 cells
  SB623 surgically implanted
- Total: Total of all reporting groups
Arm/Group | Treatment Group: 2.5 Million Cells | Treatment Group: 5 Million Cells | Treatment Group: 10 Million Cells | Sham Surgery | Total
Number analyzed (Participants) | 15 | 15 | 16 | 15 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.66 (13.57) | 31.22 (9.15) | 34.23 (11.46) | 35.48 (12.96) | 34.40 (11.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 5 | 6 | 18
  Male | 11 | 12 | 11 | 9 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 0 | 2
  Not Hispanic or Latino | 15 | 14 | 15 | 15 | 59
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 4 | 5 | 5 | 4 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 1
  White | 11 | 9 | 11 | 11 | 42
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Fugl-Meyer Motor Scale (FMMS) Score at Week 24 Among All Patients
Description: The FMMS motor component consists of the 33-item upper extremity subscale (UE-FMMS) and the 17-item lower extremity subscale (LE-FMMS). Items were scored on a 3-point ordinal scale: 0= cannot perform; 1= partial motion; 2= full motion Individual items were then summed to determine scores for the 2 subscale scores, as well as a motor total score (total of all item scores including the 2 subscales UE-FMMS and LE-FMMS). As a result, the UE-FMMS subscale score ranged from 0 to 66 and the LE-FMMS subscale score ranged from 0 to 34. The FMMS motor total score ranged from 0 (hemiplegia) to a maximum of 100 points (normal motor performance).
Time Frame: 24 weeks
Population: Modified Intent-to-Treat (mITT) Population: Included all randomized subjects who completed the surgery treatment procedure (61 subjects)
Measure: Mean (Standard Deviation); unit: Change in score on a scale from baseline
Arm/Group | Treatment Group: 2.5 Million Cells | Treatment Group: 5 Million Cells | Treatment Group: 10 Million Cells | Sham Surgery
Number analyzed (Participants) | 15 | 15 | 16 | 15
Change in score on a scale from baseline | 6.0 (10.1) | 11.0 (8.4) | 8.1 (12.8) | 2.3 (4.7)
Statistical Analysis 1: Comparison: Treatment Group: 2.5 Million Cells vs Treatment Group: 5 Million Cells vs Treatment Group: 10 Million Cells vs Sham Surgery; Adjusted LS mean and treatment group difference in change from baseline at Week 24 were modeled using an MMRM including the following variables: treatment, visit, treatment by visit interaction, baseline FMMS score, baseline FMMS score by visit interaction, GOS-E score at screening, and GOS-E score at screening by visit interaction; Test type: Superiority; p = 0.0401, Mixed Models Analysis — MMRM: Mixed Model for Repeated Measures; Least Square (LS) Mean Difference = 6.0, Standard Error of Mean 2.9

2. Secondary Outcome: Change From Baseline in Disability Rating Scale Score at Week 24 Among All Patients
Description: DRS is an observer rated, 30-point ordinal scale that evaluates eight areas of functioning in four categories:
  1. Consciousness (eye opening, verbal response, motor response)
  2. Cognitive ability (feeding, toileting, grooming)
  3. Dependence on others
  4. Employability
  Each area of functioning was rated on a scale of 0 to either 3 or 5. The maximum score is 29 (extreme vegetative state) and the minimum score is 0 (person without disability).
Time Frame: 24 weeks
Population: The Modified Intent-to-Treat (mITT) population included all randomized subjects who completed the surgery treatment procedure. Only subjects in the mITT population who have the value available for Change from Baseline in DRS at 24 weeks are included in this analysis.
Measure: Mean (Standard Deviation); unit: Change in score on a scale from baseline
Arm/Group | Treatment Group: 2.5 Million Cells | Treatment Group: 5 Million Cells | Treatment Group: 10 Million Cells | Sham Surgery
Number analyzed (Participants) | 15 | 14 | 16 | 15
Change in score on a scale from baseline | -0.1 (1.2) | -1.4 (2.6) | -0.6 (2.2) | 0.6 (1.6)
Statistical Analysis 1: Comparison: Treatment Group: 2.5 Million Cells vs Treatment Group: 5 Million Cells vs Treatment Group: 10 Million Cells vs Sham Surgery; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.1655, Mixed Models Analysis — MMRM: Mixed Model for Repeated Measures; Least Square (LS) Mean Difference = -0.7, 95% CI 2-sided [-1.7 to 0.3]

3. Secondary Outcome: Change From Baseline in ARAT Total Score at Week 24 Among Upper Extremity Deficit Patients
Description: The ARAT total score is the sum of the scores from 19 tests spread across four subscales: grasp, grip, pinch, and gross movement. Each test is scored on an ordinal 4-point scale with 0= non movement, 1 = the movement task is partially performed, 2 = the movement task is completed but takes abnormally long, and 3 = the movement is performed normally. Summation of a 0-3 score in each item yields a total score between 0 and 57.
Time Frame: 24 weeks
Population: The Modified Intent-to-Treat (mITT) population included all randomized subjects who completed the surgery treatment procedure. Only subjects in the mITT population who have the value available for Change from Baseline in ARAT at 24 weeks are included in this analysis.
Measure: Mean (Standard Deviation); unit: Change in score on a scale from baseline
Arm/Group | Treatment Group: SB623 2.5 Million Cells | Treatment Group: SB623 5 Million Cells | Treatment Group: SB623 10 Million Cells | Sham Surgery
Number analyzed (Participants) | 14 | 13 | 14 | 14
Change in score on a scale from baseline | 3.0 (6.7) | 4.2 (5.2) | -0.3 (10.3) | -0.4 (11.5)
Statistical Analysis 1: Comparison: Treatment Group: SB623 2.5 Million Cells vs Treatment Group: SB623 5 Million Cells vs Treatment Group: SB623 10 Million Cells vs Sham Surgery; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.3398, Mixed Models Analysis; MMRM included treatment, visit, baseline endpoints & GOS-E scores, baseline endpoints & GOS-E by visit interaction, treatment-by-visit interaction; Least Square (LS) Mean Difference = 2.7, 95% CI 2-sided [-2.9 to 8.3]

4. Secondary Outcome: Change From Baseline in Gait Velocity (10 Meter Walk Time in Seconds) at Week 24 Among Lower Extremity Deficit Patients
Description: Gait Velocity was measured on a standard 10 meter walk.
Time Frame: 24 weeks
Population: The Modified Intent-to-Treat (mITT) population included all randomized subjects who completed the surgery treatment procedure. Only subjects in the mITT population who have the value available for Change from Baseline in Gait Velocity at 24 weeks are included in this analysis.
Measure: Mean (Standard Deviation); unit: 10 meter walk change of time in seconds
Arm/Group | Treatment Group: SB623 2.5 Million Cells | Treatment Group: SB623 5 Million Cells | Treatment Group: SB623 10 Million Cells | Sham Surgery
Number analyzed (Participants) | 14 | 13 | 14 | 14
10 meter walk change of time in seconds | -3.1 (87.0) | -3.9 (6.7) | -2.2 (113.6) | -2.4 (6.7)
Statistical Analysis 1: Comparison: Treatment Group: SB623 2.5 Million Cells vs Treatment Group: SB623 5 Million Cells vs Treatment Group: SB623 10 Million Cells vs Sham Surgery; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.8974, Mixed Models Analysis — MMRM: Mixed Model for Repeated Measures; Least Square (LS) Mean Difference = -2.6, 95% CI 2-sided [-42.2 to 37.1]

5. Secondary Outcome: Change From Baseline in NeuroQOL T-scores at Week 24 of NeuroQOL Domains
Description: Two NeuroQoL short form assessments were used (upper extremity function and lower extremity function); each has 8 items with 5 possible scores (e.g. 1= not at all, 2=a little bit, 3= somewhat, 4=quite a bit, 5=very much) or frequency ("never"to "always"); Raw scores are converted to T-scores based on a consistent metric (i.e., the T distribution) and data from the US general population. The theoretical range in scale for Upper extremity T-score and Lower extremity T-score are 12.8 to 53.8 and 16.5 to 58.6 respectively. When interpreting these T-scores, higher scores correspond to higher levels of functioning whereas lower scores correspond to lower levels of functioning.
Time Frame: 24 weeks
Population: The Modified Intent-to-Treat (mITT) population included all randomized subjects who completed the surgery treatment procedure. Only subjects in the mITT population who have the value available for Change from Baseline in NeuroQOL T-scores at 24 weeks are included in this analysis.
Measure: Mean (Standard Deviation); unit: Change in score on a scale from baseline
Arm/Group | Treatment Group: SB623 2.5 Million Cells | Treatment Group: SB623 5 Million Cells | Treatment Group: SB623 10 Million Cells | Sham Surgery
Number analyzed (Participants) | 14 | 13 | 15 | 13
Change in score on a scale from baseline
  Change in T-score from baseline (upper extremity function) | 5.66 (8.06) | 5.27 (8.90) | -0.77 (6.42) | 2.48 (9.89)
  Change in T-score from baseline (lower extremity function) | 3.06 (6.58) | 1.95 (6.82) | 3.38 (7.10) | 1.75 (7.05)
Statistical Analysis 1: Comparison: Treatment Group: SB623 2.5 Million Cells vs Treatment Group: SB623 5 Million Cells vs Treatment Group: SB623 10 Million Cells vs Sham Surgery; Change from Baseline in NeuroQOL Upper Extremity Function T Score at Week 24; Test type: Superiority; p = 0.8534, Mixed Models Analysis — MMRM: Mixed Model for Repeated Measures; [statistical method as in outcome 3, analysis 1]; Least Square (LS) Mean Difference = -0.49, 95% CI 2-sided [-5.77 to 4.80]
Statistical Analysis 2: Comparison: Treatment Group: SB623 2.5 Million Cells vs Treatment Group: SB623 5 Million Cells vs Treatment Group: SB623 10 Million Cells vs Sham Surgery; Change from Baseline in NeuroQOL Lower Extremity Function T Score at Week 24; Test type: Superiority; p = 0.8443, Mixed Models Analysis — MMRM: Mixed Model for Repeated Measures; [statistical method as in outcome 3, analysis 1]; Least Square (LS) Mean Difference = 0.41, 95% CI 2-sided [-3.78 to 4.60]

6. Secondary Outcome: Global Rating of Perceived Change: The Percentage of Subjects Scoring Either 6 or 7 on the Global Rating of Perceived Change by Both Subject and Physician
Description: The proportions of SB623 treated subjects (pooling all SB623 doses) scoring either 7 (much better) or 6 (a little better, meaningful) on the Global Rating of Perceived Change (from Baseline) - Subject at Week 24 and on the Global Rating of Perceived Change (from Baseline) - Clinician at Week 24 was compared to the corresponding proportions of sham surgery control subjects using logistic regression models with adjustment for the baseline Fugl-Meyer Motor Scale score and the GOS-E score at screening as continuous covariates. The following 7-point Likert scale was used
  * Score 7 = Much better
  * Score 6 = A little better, meaningful
  * Score 5 = A little better, not meaningful
  * Score 4 = About the same
  * Score 3 = A little worse, not meaningful
  * Score 2 = A little worse, meaningful
  * Score 1 = Much worse
Time Frame: 24 weeks
Population: Modified Intent-to-Treat (mITT) Population: Included all randomized subjects who completed the surgery treatment procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group: SB623 2.5 Million Cells | Treatment Group: SB623 5 Million Cells | Treatment Group: SB623 10 Million Cells | Sham Surgery
Number analyzed (Participants) | 15 | 15 | 16 | 15
Participants
  Clinician at Week 24: Scoring either 6 or 7 on the Global Rating (Yes) | 5 | 6 | 4 | 2
  Clinician at Week 24: Scoring either 6 or 7 on the Global Rating (No) | 10 | 9 | 12 | 13
  Subject at Week 24: Scoring either 6 or 7 on the Global Rating (Yes) | 8 | 12 | 6 | 4
  Subject at Week 24: Scoring either 6 or 7 on the Global Rating (No) | 7 | 3 | 10 | 11

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Treatment Group: SB623 2.5 Million Cells | Treatment Group: SB623 5 Million Cells | Treatment Group: SB623 10 Million Cells | Sham Surgery
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/16 | 0/15
Serious Adverse Events (participants affected / at risk) | 1/15 | 1/15 | 2/16 | 3/15
Other Adverse Events (participants affected / at risk) | 15/15 | 15/15 | 16/16 | 14/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Group: SB623 2.5 Million Cells (N=15) | Treatment Group: SB623 5 Million Cells (N=15) | Treatment Group: SB623 10 Million Cells (N=16) | Sham Surgery (N=15)
Wound infection (Infections and infestations) | 0 | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Balance disorder (Nervous system disorders) | 0 | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 0 | 1 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Group: SB623 2.5 Million Cells (N=15) | Treatment Group: SB623 5 Million Cells (N=15) | Treatment Group: SB623 10 Million Cells (N=16) | Sham Surgery (N=15)
Headache (Nervous system disorders) | 5 | 6 | 8 | 4
Wound complication (Injury, poisoning and procedural complications) | 3 | 5 | 4 | 3
Nausea (Gastrointestinal disorders) | 3 | 3 | 2 | 1
Vomiting (Gastrointestinal disorders) | 2 | 2 | 4 | 1
Pyrexia (General disorders) | 4 | 2 | 0 | 0
Asthenia (General disorders) | 2 | 2 | 1 | 1
Dizziness (Nervous system disorders) | 3 | 1 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 2
Incision site pain (Injury, poisoning and procedural complications) | 3 | 0 | 1 | 1
Procedural headache (Injury, poisoning and procedural complications) | 2 | 0 | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 3 | 1 | 0
Agitation (Psychiatric disorders) | 2 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 2 | 0
Head discomfort (Nervous system disorders) | 1 | 1 | 1 | 0
Influenza (Infections and infestations) | 1 | 0 | 2 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-05-17): https://cdn.clinicaltrials.gov/large-docs/92/NCT02416492/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-16): https://cdn.clinicaltrials.gov/large-docs/92/NCT02416492/SAP_001.pdf